CLINICAL TRIAL: NCT02983721
Title: Comparison Between Transradial and Transfemoral Routes of Coronary Angiography and Interventions
Brief Title: Trans Radial Versus Transfemoral Route for Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheri Kashmir Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Khalid Changal, Principal Investigator, Sheri Kashmir Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: car003421; PG thesis 003421 (Other: Sher-i-Kashmir Institute of Medical Sciences)
Record Dates: First submitted 2016-12-01; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transfemoral (Active Comparator): in case of transfemoral approach our preference was to use right femoral route. The groin was prepared and draped and the site was punctured for femoral access after anesthetizing the skin with 2-4 ml of 1% lignocaine. Once the femoral puncture was done 6F sheath of Cordis variety was introduced and 6F Judkins, catheter was introduced and it was guided under fluoroscopic guidance through the aortic route.
  Interventions: Procedure: transradial; Procedure: Transfemoral
- Transradial (Active Comparator): Our preference was to use the right radial and right femoral routes as they are nearest to operator while facing cardiac monitors, in our hospital. For the radial approach, the wrist was sterilized and draped in usual fashion. Hyperextension over an arm board was done and skin over the puncture site was anesthetized with 2 - 3 ml of 1% lignocaine. A small scaled incision was performed 1 cm proximal to styloid process of radius where arterial pulse was best felt. The radial artery was punctured with a 21 G needle and 6 F sheath (Cardis, Terumo) were introduced into the artery, using Seldinger technique. All patients received verapamil (5mg) to reduce radial artery spasm. Heparin (weight adjusted) was used only in PCIs to prevent artery occlusion and not in elective diagnostic coronary studies. Long 0.038 Terumo guide wire was used under fluoroscopic guidance.
  Interventions: Procedure: transradial; Procedure: Transfemoral

INTERVENTIONS:
Procedure: transradial — transradial route for coronary angiography and PCI
Procedure: Transfemoral — transfemoral route for coronary angiography and PCI

SUMMARY:
The purpose of this study was to assess and compare the feasibility, success and safety of Transradial approach (TRA) verses Transfemoral approach (TFA) for diagnostic and therapeutic coronary angiography and coronary interventions, in terms of procedural time, access time, fluoroscopy time, procedural failure, , length of hospital stay in terms of days in hospital, Complications in terms of thrombophlebitis, hematoma, ecchymosis, infections thrombosis of vessel, MACE, Stroke and others.

DETAILED DESCRIPTION:
Background: PCI has been done traditionally through transfemoral route. But now transradial and transbrachial routes are also coming up in practice. We compared transradial versus transfemoral routes for ease of operability, time for procedure, complications, and failure rates through a prospective study. Methods: 400 Patients admitted in department of cardiology for percutaneous interventions were enrolled in the study. 200 patients were assigned to each group randomly. A single team did all the procedures. Pre procedure, intra procedure and post procedure data of all the patients was collected, tabulated and analysed properly.

The variables studied include Access time ,Fluoroscopy time and overall procedure time, post procedure complications( ecchymosis ,Thrombophelibites, Hematoma, procedure access bleed), Failure rates,post procedure myocardial infarction, stroke, acute renal failure and infections.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic angiography of coronary vessels, PCI

Exclusion Criteria:

* Patients with impaired renal function tests.

  * Lack of informed consent.
  * Severe infection.
  * Previous contrast allergy.
  * Severe intrinsic/iatrogenic caogulopathy INR>2.
  * Abnormal modified Allen's test.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Access time | 4 years
  Access time for the procedures
Fluoroscopy time | 4 years
  measure of radiation exposure
Procedure time | 4 years
  time taken to do the full procedure
hospital stay | 4 years
  time period the patient stayed in the hospital

SECONDARY OUTCOMES:
hematoma | 4 years
  hematoma development at the site of puncture
pseudoaneurysm | 4 years
  local complication at the access site
bleeding | 4 years
  at the access site
Access site failure | 4 years
  failure to gain access for the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fayaz Bhat, MBBS, MD, Study Chair — Ministry of Health, Jammu and Kashmir, India.

IPD SHARING:
Plan to Share IPD: Yes
can be shared by email

REFERENCES:
- [Derived] Bhat FA, Changal KH, Raina H, Tramboo NA, Rather HA. Transradial versus transfemoral approach for coronary angiography and angioplasty - A prospective, randomized comparison. BMC Cardiovasc Disord. 2017 Jan 11;17(1):23. doi: 10.1186/s12872-016-0457-2. PMID 28077091